CLINICAL TRIAL: NCT02684864
Title: Does the Biological Response to Degenerative Meniscal Tears or to Their Intervention Predict Future Osteoarthritis?: The Meniscal Tear and Osteoarthritis Risk (MenTOR) Study
Brief Title: Meniscal Tear and Osteoarthritis Risk (MenTOR)
Acronym: MenTOR
Status: Active, not recruiting | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: Oxford University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: PID 11499
Record Dates: First submitted 2016-01-20; First posted 2016-02-18 (Estimated); Last update posted 2021-04-01 (Actual); Status verified 2020-11

CONDITIONS: Osteoarthritis
Keywords: biomarker; inflammation; knee; prognosis
MeSH Terms: conditions — Osteoarthritis; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples (plasma, serum, DNA where consent is given), urine, synovial fluid (where an appropriate clinically indicated procedure has been carried out to allow access).
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Non-interventional

SUMMARY:
Adults with degenerative meniscal tear receiving arthroscopic surgical management or knee drainage (arthrocentesis) +/- intra-articular steroid injection will be recruited to this non-interventional cohort study. The aim is to investigate whether measurement of an individual's synovial fluid biomarker response to a degenerative meniscal tear with symptoms predicts symptomatic and functional outcome suggestive of osteoarthritis (OA) of the knee.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 30-60 years.
2. Participant able and willing to give informed consent.
3. Clinical assessment demonstrates mechanical symptoms suggestive of meniscal pathology (focal knee pain +/- 1 or more of: catching/locking, giving way, focal joint-line tenderness, effusion, McMurray's positive) within last 12 months.
4. Evidence on clinical MRI knee of meniscal tear.
5. Participant is either in secondary care or has the potential to be referred to secondary care due to severity of symptoms.
6. Patient has failed conservative therapy and elected for surgical arthroscopic treatment, or is due knee drainage/injection for clinical reasons.
7. Competency of the English language to complete questionnaires independently.

Exclusion Criteria:

1. Pre-existing advanced radiographic OA (KL grade 3-4) of index knee at baseline.
2. Evidence of anterior cruciate ligament rupture, or more extensive soft tissue injury.
3. History of an acute knee injury (within 12 weeks), or acutely locked knee
4. Known history of inflammatory/septic arthritis of index knee.
5. Knee replacement or other non-arthroscopic knee surgery (e.g. high tibial osteotomy) - previous or planned within 1 year of study start.
6. Index knee surgery within last 3 months, including meniscectomy.
7. Steroid injection to index knee in last 3 months.
8. Active other (treated) inflammatory disease or infection.
9. Positive pregnancy test.
10. Unable to provide blood samples.
11. Unable to give informed written consent.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with a confirmed meniscal tear, likely degenerative in nature, will be invited to participate in the MenTOR study. Male and female adults with a MRI-evident meniscal tear and evidence of no/minor osteoarthritic change (KL grade 2 or less) who are undergoing arthroscopic treatment, or planned arthrocentesis/injection will be identified in clinics all located at the Nuffield Orthopaedic Centre (NOC). The primary source of recruitment is anticipated to be the secondary care orthopaedic knee service. The patient's symptoms will be such that they warrant further management.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2016-03 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Knee Injury and Osteoarthritis Outcomes Score (KOOS)-4 | 2 years
  summary score from validated KOOS questionnaire. To investigate whether measurement of an individual's synovial fluid biomarker response to a degenerative meniscal tear with symptoms predicts symptomatic and functional outcome suggestive of OA of the knee.

SECONDARY OUTCOMES:
X ray Kellgren Lawrence (KL) change | 2 years
  X ray of knee.Change in KL grade over time will be measured.
MRI semi-quantitative score | 2 years
  MRI knee. Change in semi-quantitative score over time will be measured.
Oxford Knee Score - Activity and Participation Questionnaire (OKS-APQ) | 2 years
  The OKS-APQ will be used to document pain and symptoms, and compared with KOOS.

CONTACTS AND LOCATIONS:
Overall Officials: Fiona Watt, MD, PhD, Principal Investigator — University of Oxford
Locations (1):
- Kennedy Insitute of Rheumatololgy, NDORMS, University of Oxford, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: OA centre homepage — http://oacentre.kennedy.ox.ac.uk/